CLINICAL TRIAL: NCT06093061
Title: RIBBON-LA-01: Single-arm, Open-label, Phase 2 Trial of Tislelizumab and Metronomic Capecitabine as Maintenance Therapy in High-risk Locoregionally-advanced Nasopharyngeal Carcinoma
Brief Title: Tislelizumab and Metronomic Capecitabine as Maintenance in High-risk Locoregionally-advanced Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: BeiGene (Industry); Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIBBON-LA-01
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Locoregionally-advanced NPC; EBV DNA; Concurrent chemoradiotherapy (CCRT); Maintenance Tislelizumab; Metronomic Capecitabine
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAINTENANCE STUDY TREATMENT (Experimental): EBV DNA ≥4000 copies/mL OR N3 OR T4N+ (TNM AJCC/UICC 8th edition) AND EBV DNA detectable after 3 cycles of IC.
  Interventions: Combination Product: CCRT with Maintenance Tislelizumab and Metronomic Capecitabine

INTERVENTIONS:
Combination Product: CCRT with Maintenance Tislelizumab and Metronomic Capecitabine — CCRT: Radiotherapy will be delivered once daily, for 5 days per week, over 6 to 7 weeks. During RT, cisplatin will be administered either 100 mg/m2 3-weekly or 40 mg/m2 weekly, IV infusion (physician's choice).
  Maintenance: Tislelizumab 200mg, day 1 per 3-week cycle, intravenous (IV) infusion and capecitabine 650 mg/m2, days 1-21 per 3-week cycle, bidaily, oral, for a total of 12 months (17 cycles).

SUMMARY:
Patients with "high-risk" locoregionally-advanced nasopharyngeal carcinoma (LA-NPC), defined as AJCC/UICC 8th edition TNM-stage III-IVA and high Epstein-Barr virus (EBV) DNA viral load (≥4,000 copies/mL) will require induction chemotherapy (IC) prior to chemo-radiation (CCRT) as per standard treatment. Patients who persist to manifest DETECTABLE EBV DNA following 3 cycles of IC have a higher risk of relapse, and are typically recommended for a year of low-dose oral chemotherapy after CCRT.

RIBBON-LA-01 is a single-arm, open-label, phase 2 clinical trial of maintenance tislelizumab and metronomic capecitabine (metroCap) for 52 weeks after IC and CCRT, targeting this specific group of patients who have persistent detectable EBV DNA after IC. The main objective is to evaluate the efficacy of maintenance tislelizumab and metroCap in patients with DETECTABLE EBV DNA levels after 3 cycles of IC.

DETAILED DESCRIPTION:
RIBBON-LA-01 is embedded in a modular platform trial concept (NCT05517135, https://clinicaltrials.gov/study/NCT05517135) that tests if EBV DNA-based risk stratification strategies for treatment individualization improves survival outcomes in LA-NPC. The overarching platform trial concept allocates patients with LA-NPC to treatment arms of different intensities by their plasma EBV DNA levels pre-treatment and post-IC.

RIBBON-LA-01 enrolls patients allocated to Arm 3 of the platform trial; these are patients with pre-treatment EBV DNA of >4,000 copies/mL OR N2-3 or T4N+ NPC who were treated with upfront IC, but persist to manifest DETECTABLE EBV DNA levels following 3 cycles of IC. Patients on the trial will be assigned to CCRT followed by a 12-month course of maintenance tislelizumab and metroCap.

The primary endpoint of the study is two-year disease free survival, defined as the proportion of patients who are alive and free of disease relapse at the end of 2 years after the start of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments
2. Age ≥21 years on the day of signing the ICF
3. ECOG Performance Status ≤1
4. Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and ≥120 days after the last dose of tislelizumab, and have a negative urine or serum pregnancy test ≤7 days of start of trial
5. Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study and for ≥120 days after the last dose of tislelizumab

Exclusion Criteria:

1. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137)
2. Has received any prior radiotherapy (RT) or systemic anti-cancer therapy including investigational agents for NPC
3. Any known central nervous system metastases and/or carcinomatous meningitis
4. Active autoimmune diseases or history of autoimmune diseases that may relapse

   Note: Patients with the following diseases are not excluded and may proceed to further screening:
   1. Controlled Type I diabetes
   2. Hypothyroidism (provided it is managed with hormone replacement therapy only)
   3. Controlled celiac disease
   4. Skin diseases not requiring systemic treatment (e.g., vitiligo, psoriasis, alopecia)
   5. Any other disease that is not expected to recur in the absence of external triggering factors
5. Any active malignancy ≤2 years before start of study except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively (e.g., resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast)
6. Any condition that required systemic treatment with either corticosteroids (>10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤14 days before start of study

   Note: Patients who are currently or have previously been on any of the following steroid regimens are not excluded:
   1. Adrenal replacement steroid (dose ≤10 mg daily of prednisone or equivalent)
   2. Topical, ocular, intra-articular, intranasal, or inhaled corticosteroid with minimal systemic absorption
   3. Short course (≤7 days) of corticosteroid prescribed prophylactically (e.g., for contrast dye allergy) or for the treatment of a non-autoimmune condition (e.g., delayed-type hypersensitivity reaction caused by contact allergen)
7. With uncontrolled diabetes or >Grade 1 laboratory test abnormalities in potassium, sodium, or corrected calcium despite standard medical management or ≥Grade 3 hypoalbuminemia ≤14 days before start of study
8. With history of interstitial lung disease, non-infectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases, etc.
9. With severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection, etc.

   1. Severe infections within 4 weeks before start of study, including but not limited to hospitalization for complications of infection, bactiraemia, or severe pneumonia.
   2. Received therapeutic oral or intravenous antibiotics within 2 weeks before start of study.
10. A known history of HIV infection
11. Patients with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers whose HBV DNA is >500 IU/mL or patients with active hepatitis C virus (HCV) should be excluded. Note: Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B (HBV DNA <500 IU/mL), and cured hepatitis C patients can be enrolled
12. Any major surgical procedure requiring general anaesthesia ≤28 days before start of study
13. Prior allogeneic stem cell transplantation or organ transplantation
14. Any of the following cardiovascular risk factors:

    1. Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, ≤28 days before start of study
    2. Pulmonary embolism ≤28 days before start of study
    3. Any history of acute myocardial infarction ≤6 months before start of study
    4. Any history of heart failure meeting New York Heart Association (NYHA) Classification III or IV ≤6 months before start of study
    5. Any event of ventricular arrhythmia ≥Grade 2 in severity ≤6 months before start of study
    6. Any history of cerebrovascular accident ≤6 months before start of study
    7. Uncontrolled hypertension: systolic pressure ≥160 mmHg or diastolic pressure ≥100 mmHg despite anti-hypertension medications ≤28 days before start of study
    8. Any episode of syncope or seizure ≤28 days before start of study
15. A history of severe hypersensitivity reactions to tislelizumab, gemcitabine, cisplatin, capecitabine and/or any of its excipients
16. Has received any herbal medicine used to control cancer within 14 days of the start of study
17. Patients with toxicities (as a result of prior anticancer therapy) which have not recovered to baseline or stabilized, except for AEs not considered a likely safety risk (e.g., alopecia, neuropathy and specific laboratory abnormalities)
18. Was administered a live vaccine ≤4 weeks before start of study Note: Seasonal vaccines for influenza are generally inactivated vaccines and are allowed. Intranasal vaccines are live vaccines, and are not allowed
19. Underlying medical conditions (including laboratory abnormalities) or alcohol or drug abuse or dependence that, will be unfavourable for the administration of study drug or affect the explanation of drug toxicity or AEs or result in insufficient or might impair compliance with study conduct
20. Concurrent participation in another therapeutic clinical study

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
2-year Disease-Free Survival (DFS) rate. | 2 Years.
  The proportion of patients who are alive and free of disease relapse at the end of 2 years after the start of Induction Chemotherapy (IC) for patients.

SECONDARY OUTCOMES:
3-year Overall Survival (OS). | 3 years.
  Time from date of start of treatment (IC) to death from any cause, where patients lost to follow-up were censored at the date of last follow-up.
Distant Metastasis-Free Survival (DMFS). | 2 years.
  Time from date of start of treatment (IC) to documented distant metastasis or death from any cause, patients with locoregional relapse as a first event will be censored at date of locoregional relapse
Loco-Regional Recurrence-Free Survival (LRRFS). | 2 years.
  Time from date start of treatment (IC) to documented locoregional relapse or death from any cause, patients with distant metastasis as a first event will be censored at the date of distant metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Melvin LK CHUA, MBBS, FRCR, PhD, FAMS, Principal Investigator — National Cancer Centre, Singapore
Locations (2):
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Yes
With BeiGene.